CLINICAL TRIAL: NCT04348084
Title: Oncologic Impact of Pancreatic Fistula After Distal Pancreatectomy for Pancratic Ductal Adenocarcinoma oh the Body and the Tail : a Multicentre Retrospective Cohort Analysis / POPF-DSS (Postoperative Pancreatic Fistula - Disease Specific Survival)
Brief Title: Oncologic Impact of Pancreatic Fistula
Acronym: POPF-DSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: IRCCS San Raffaele (Other); Cisanello University Hospital (Pisa, Italy) (Unknown); Reims University Hospital (Reims, France) (Unknown); Rennes University Hospital, Rennes, France (Unknown); Morgagni Pierantoni Hospital (Other); Fondazione Poliambulanza Hospital (Brescia, Italy) (Unknown); Grenoble Alpes University Hospital (Grenoble, France) (Unknown); SS. Antonio e Biagio e Cesare Arrigo Hospital (Alessandria, Italy) (Unknown); University of Bari (Other); IHU Strasbourg (Strasbourg, France) (Unknown); Hospital Centre of Luxemburg (Luxemburg) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0213
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: PDAC of the Body and the Tail of the Pancreas; CR- POPF
Keywords: Clinically relevant pancreatic fistula; pancreatic leak; pancreatic cancer; left pancreatectomy; distal pancreatectomy; oncologic outcome; pancreatic cancer recurrence
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- who developed POPF: Patients undergone curative distal pancreatectomy for PDAC who developed POPF
- who did not develop POPF: Patients undergone curative distal pancreatectomy for PDAC who did not develop POPF

SUMMARY:
Clinically-relevant post-operative fistula is a major complication after DP, but it did not affect post-operative therapeutic path nor oncologic long-term outcomes. CR-POPF was not a predictive factor for disease recurrence and it was not associated with an increased incidence of peritoneal or local relapse.

DETAILED DESCRIPTION:
POPF is the most common and feared complication after distal pancreatectomy (DP), increasing morbidity and mortality. Recent evidences suggest that POPF can also play a role in pancreatic cancer recurrence. Adult patients with a diagnosis of pancreatic ductal adenocarcinoma (PDAC) of the body and tail of the pancreas, undergoing curative DP, over a ten-year period in twelve European Surgical Departments were retrospectively collected from a prospective implemented database. Cohort studied included 283 patients, 139 were men (49.1%), median age was 70 years-old (range 37-88). A total of 121 POPF were observed (42.8%), 42 of them (14.9%) were CR-POPF. Median follow-up period was 24 months (range 3-120). Although poorer in the POPF group, overall survival (OS) and disease-free survival (DFS) did not differ significantly when comparing patients with and without CR-POPF (p= 0.224 and p= 0.165, respectively). CR-POPF was not significantly associated with local or peritoneal recurrence (p=0.559 and p=0.302, respectively). Less patients after POPF (76.2% versus 83.8%) benefited from adjuvant chemotherapy but the difference was not significant (p=0.228). CR-POPF is a major complication after DP, but it did affect neither the post-operative therapeutic path nor oncologic outcomes. CR-POPF was not a predictive factor for disease recurrence and it was not associated with an increased incidence of peritoneal or local relapse.

ELIGIBILITY:
Inclusion criteria:

- patient with resectable pancreatic ductal adenocarcinoma (PDAC) of the body and the tail of the pancreas undergone surgery

Exclusion criteria:

* metastatic diseases (including para-aortic lymph nodes involvement)
* PDAC arising from Intraductal Papillary Mucinous Neoplasms (IPMN)
* resection for premalignant lesions including high-grade Pancreatic Intraepithelial Neoplasia (PanIN) or adenocarcinoma in situ (Tis)
* histological diagnosis other than PDAC
* all R2 resections.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with a diagnosis of pancreatic ductal adenocarcinoma (PDAC) of the body and the tail of the pancreas, undergoing DP with curative intent, over a ten-year period (from January 2009 to December 2018) in twelve European Surgical Departments were retrospectively collected from a prospective implemented database.
Sampling Method: Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2009-01-30 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
impact of clinically relevant (CR-) POPF | 10 years
  The primary aim of this study is to assess the impact of clinically relevant (CR-) POPF on patient disease specific survival (OS and DFS) after curative distal pancreatectomy.

SECONDARY OUTCOMES:
identifying positive and negative prognostic factors | 10 years
  Secondary end-points of the analysis are aimed at identifying positive and negative prognostic factors and at investigating the role of POPF in specific site recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio PANARO, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Leon P, Giannone F, Belfiori G, Falconi M, Crippa S, Boggi U, Menonna F, Al Sadairi AR, Piardi T, Sulpice L, Gardini A, Sega V, Chirica M, Ravazzoni F, Giannandrea G, Pessaux P, de Blasi V, Navarro F, Panaro F. The Oncologic Impact of Pancreatic Fistula After Distal Pancreatectomy for Pancreatic Ductal Adenocarcinoma of the Body and the Tail: A Multicenter Retrospective Cohort Analysis. Ann Surg Oncol. 2021 Jun;28(6):3171-3183. doi: 10.1245/s10434-020-09310-y. Epub 2020 Nov 6. PMID 33156465